CLINICAL TRIAL: NCT03677453
Title: Interactive Perioperative Teaching Platform (IPTP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Associate Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB17-01340
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Tonsillar Hypertrophy; Adenoid Hypertrophy; Cryptorchidism; Hypospadias; Hydrocele
MeSH Terms: conditions — Cryptorchidism; Hypospadias; Testicular Hydrocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPTP (Active Comparator): Patients will have access to the web-based interactive teaching tool.
  Interventions: Other: Interactive Perioperative Teaching Platform
- Non-IPTP (No Intervention): Patients will not have access to the web-based interactive teaching tool.

INTERVENTIONS:
Other: Interactive Perioperative Teaching Platform — An active video format will be used to provide instructions for navigating the hospital; describe induction of anesthesia and the surgical procedure; and provide post-surgery and post-discharge instructions for pain management.
  Other Names: IPTP
  Arms: IPTP

SUMMARY:
The proposed study will assess whether an interactive perioperative teaching platform (IPTP) provided to families of patients undergoing ambulatory pediatric surgery will reduce families' anxiety, and improve satisfaction and understanding, relative to current practice. The IPTP will educate patient families on the continuum of their child's surgical experience, from arriving at the hospital through registration, the operating room (OR), and the hospital floor. An active video format will be used to provide instructions for navigating the hospital; describe induction of anesthesia and the surgical procedure; and provide post-surgery and post-discharge instructions for pain management. A comparison cohort of patients undergoing surgery without access to the IPTP will be recruited to assess the benefits of the IPTP for improving metrics of family satisfaction, preoperative anxiety, and postoperative understanding of discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years
* Undergoing adenotonsillectomy or orchiopexy, hydrocele or hypospadias repair
* Only patients booked for ambulatory surgery in the main operating room (OR)

Exclusion Criteria:

* Patients will be excluded if they have previously undergone surgery or require a translator

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Patient family satisfaction | Immediately prior to discharge
  Family satisfaction will be assessed by a member of the research team using an adaptation of the English version of the Leiden Perioperative Patient Satisfaction questionnaire (LPPSq) recommended for research on satisfaction with surgeries involving anesthesia. The English version assesses 4 domains of satisfaction: information provision, professional competence, patient-staff relationship, and service with a total of 24 questions on these topics. It is scored on a 1-5 Likert scale (from completely dissatisfied to completely satisfied).

SECONDARY OUTCOMES:
Anxiety level | Baseline
  Anxiety will be measured using the short-form State-Trait Anxiety Inventory 10 with scores ranging from 6-24 (least to most anxious).

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No